CLINICAL TRIAL: NCT04958278
Title: Pelvic Sentinel Node According to SHREC-trial for the Application of the 2021 European Recommendations for Lymph Node Staging Strategy in Endometrial Cancer
Brief Title: Pelvic Sentinel Node Detection Using Indocyanine Green Learning Curve
Acronym: ENDO-GREEN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ENDO-GREEN ( 29BRC21.0078)
Record Dates: First submitted 2021-07-01; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-04

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to ESGO-ESTRO-ESMO guidelines, pelvic Sentinel lymph node detection is suitable for lymph node staging in endometrial carcinoma of the uteri.

Nonetheless, a learning curve is mandatory to ensure the surgical quality of the sampling.

The aim of the study is to assess the success of sentinel lymph node detection according to SHREC-Trial surgical strategy.

DETAILED DESCRIPTION:
Introduction:

According to ESGO-ESTRO-ESMO guidelines, pelvic Sentinel lymph node detection is suitable for lymph node staging in endometrial carcinoma of the uteri.

The aim of the study is to assess the success of sentinel lymph node detection according to SHREC-Trial surgical strategy.

Patients and Method:

All patients presenting with early FIGO stage and low, intermediate, high intermediate or high risk endometrial carcinoma will be prospectively enrolled.

Sentinel lymph node mapping will be performed using laparoscopic approach and cervical Indocyanine Green injection.

Based on the surgical algorithm for detection of pelvic sentinel lymph node in endometrial cancer from Persson and coll., we designed a study with a target of 70% to 90% of bilateral detection rate .

Thirty patients will be included over 18 months.

ELIGIBILITY:
Inclusion Criteria:

Letter of non objection Endometrial carcinoma Stage FIGO I-II whatever the histological subtype. ESGO-ESMO-ESTRO 2021 risk classification : low, intermediate, high intermediate, high Laparoscopic approach.

Exclusion Criteria:

Participation refusal Medical contraindication to laparoscopic approach. Stage FIGO > II Suspected Indocyanine Green allergy

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: 30 patients over 18 months total duration of the study 20 months
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Bilateral node detection rates | Day 0 (during surgery)
  target = 70% to 90%

SECONDARY OUTCOMES:
sentinel nodes | Day 0 (during surgery)
  number of sentinel nodes collected
Salvage operations in case of GS failure | Day 0 (during surgery)
  Number of salvage operations
adverse events | Day 30
  Per and post operative adverse events according to Clavine Dindo Classification
factors for detection failure | Day 0 (during surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 18 month and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.